CLINICAL TRIAL: NCT01601119
Title: The Impact of Disease Modifying Therapies (DMTs) and Associated Support Services on Patient Reported Experience Measures (PREMs) and Outcomes (PROs) in Relapsing Multiple Sclerosis (RMS) Patients
Brief Title: Impact of Disease Modifying Therapies (DMTs) and Associated Support Services in Relapsing Multiple Sclerosis (RMS) Patients
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Limited, UK (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR200136_550
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: Multiple Sclerosis; Patient reported outcome; Patient reported experience
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Rebif cohort: Subject will receive Rebif as the treatment medication as per the standard or current practices or as directed by the healthcare professional. Allocation of subjects to a specific cohort was based on the first DMT they will be prescribed regardless of any subsequent treatment switches.
  Interventions: Drug: Rebif
- Other DMT cohort: Subjects will receive DMT other than Rebif as per the standard or current practices or as directed by the healthcare professional. Allocation of subjects to a specific cohort was based on the first DMT they will be prescribed regardless of any subsequent treatment switches.
  Interventions: Other: Other: Disease modifying therapies (DMT)

INTERVENTIONS:
Drug: Rebif — The subjects will receive Rebif as per the current practices or as directed by the physician.
  Groups: Rebif cohort
Other: Other: Disease modifying therapies (DMT) — The subjects will receive other DMTs as per the current practices or as directed by the physician.
  Groups: Other DMT cohort

SUMMARY:
The objective is to establish the impact of current disease modifying therapies (DMTs) and associated support services on Patient Reported Experience Measures and Patient Reported Outcomes in relation to the treatment and management of Relapsing Multiple Sclerosis in the United Kingdom (UK).

ELIGIBILITY:
Inclusion Criteria:

* Relapsing Multiple Sclerosis patients aged 18 years or over.
* Naive to previous DMT therapy and not yet started treatment with a disease modifying therapy.

Exclusion Criteria:

* Participating in an MS-related clinical trial.
* Unwilling to provide electronic online consent.
* Any disability that may impair them from being able to complete the online questionnaire.
* Do not have regular access to the Internet.
* Unable to complete the baseline questionnaire before they receive their first DMT injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the UK newly diagnosed with RMS (and naive to previous DMT) and receiving a DMT that can be self-administered
Sampling Method: Non-Probability Sample
Enrollment: 545 (Actual)
Dates: Start 2012-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Treatment Satisfaction | 96 weeks
  The survey sample size has been calculated based on the TSQM-9 questionnaire in order to compare scores between both patient cohorts.

SECONDARY OUTCOMES:
Work Productivity | 96 weeks
  Work Productivity and Activity Impairment (WPAI) Questionnaire
Health Related Quality of Life | 96 weeks
  Multiple Sclerosis Impact Scale (MSIS-29) v2.0 Questionnaire
Health Related Quality of Life EuroQoL (EQ-5D)-5L Questionnaire | 96 weeks
Device satisfaction | 96 weeks
  Multiple Sclerosis Treatment Concerns Questionnaire (MSTCQ) is an MS-specific treatment satisfaction questionnaire that evaluates injection system satisfaction and side effects.
Evaluation of support services | 96 weeks
  Patient evaluation of Manufacturer, Homecare and NHS support services

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Serono Limited, UK
Locations (1):
- Please contact the, Merck KGaA Communication Center For Locations, United Kingdom